CLINICAL TRIAL: NCT04647123
Title: Evaluation of Ischemic Modified Albumin, Catalase, Reduced Glutathione, Malondialdehyde, Adenosine Deaminase Levels in Blood, Saliva and Gingival Fluid in Periodontitis
Brief Title: Evaluation of Biomarker Levels in Blood, Saliva and Gingival Fluid in Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacer Sahin Aydinyurt, Assoc. Prof., Yuzuncu Yil University
Other Study IDs: : 06.06.2018/09
Record Dates: First submitted 2020-11-17; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Periodontitis
Keywords: periodontitis; catalase; malondialdehide
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hopeless teeth: The teeth that can not be treated periodontally and who are desperate for extraction will be included in this group.
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (hopeless, periodontitis, gingivitis, healthy)
- Periodontitis: Teeth diagnosed with periodontitis will be included in this group.
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (hopeless, periodontitis, gingivitis, healthy)
- Gingivitis: Teeth diagnosed with gingivitis will be included in this group.
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (hopeless, periodontitis, gingivitis, healthy)
- Healthy: Teeth diagnosed with helthy will be included in this group.
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (hopeless, periodontitis, gingivitis, healthy)

INTERVENTIONS:
Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis (hopeless, periodontitis, gingivitis, healthy) — No intervention was applied to the groups the samples will be collected in terms of the diagnosis (hopeless, periodontitis, gingivitis, healthy)

SUMMARY:
The aim of this study was to compare IMA, MDA, CAT, GSH and ADA levels in gingival crevicular fluid, serum and saliva of periodontally hopeless, periodontitis and gingivitis teeth with healthy control groups.

DETAILED DESCRIPTION:
The research methodology was approved by the Van Yuzuncu Yıl University Clinical Research Ethics Committee. (Decision number: 06.06.2018/09).

The aim of this study is to compare Ischemia-modified albumin (IMA), malondialdehyde (MDA), Catalase (CAT), Glutathione (GSH) and Adenosine deaminase (ADA) levels in gingival crevicular fluid, serum and saliva of periodontally hopeless, periodontitis and gingivitis teeth with healthy control groups.

In this study, 25 periodontally healthy individuals (control group) and 25 individuals with various levels of periodontal disease in different teeth will be included.

Gingival crevicular fluid, saliva and blood samples will be taken from patients with periodontally healthy teeth without any treatment.

In patients diagnosed with periodontal disease, teeth will be divided into 3 subgroups as hopeless, periodontitis and gingivitis. In patients with a diagnosis of periodontal disease, saliva and blood samples will be taken twice, before and after the training of scaling and root planing, desperate tooth extraction, oral hygiene motivation.

ELIGIBILITY:
Inclusion Criteria:

Systemically healhty non-smokers non-pregnants -

Exclusion Criteria:

- Patients with systemic disease smokers pregnants

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Systemically healhty ,non-smokers,non-pregnants will be included in the study
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
adenosine deaminase | 1 year
  Adenosine deaminase (ADA) is an enzyme involved in proliferation and differentiation. Although ADA has been investigated in different inflammatory and infectious diseases and has been defined as an immunoenzyme biomarker, its role in periodontitis has not been fully elucidated yet.
catalase | 1 year
  Catalase (CAT) decomposes H2O2 catalyzed by superoxide dismutase (SOD) into H2O and O2. (13) It is stated in the literature that CAT, SOD and total oxidant state are important biomarkers that can be used in the diagnosis of periodontal disease and evaluation of treatment results. (14)
Ischemia-modified albumin | 1 year
  Ischemia-modified albumin (IMA) is suggested as an oxidative stress marker and an indicator of inflammatory diseases. It has been reported in the literature that the serum IMA level increases significantly in the case of periodontal disease and decreases after treatment. In this respect, it has been stated that IMA can be an indicator of systemic inflammation caused by periodontal disease.
malondialdehide | 1 year
  In periodontal disease, an increase in reactive oxygen species and a decrease in antioxidant activity are observed because this disease is thought to be associated with an imbalance between antioxidants and oxidants. (8) Lipid peroxidation is a result of periodontitis. Free radicals that lead to the production of toxic and reactive aldehyde metabolites such as malondialdehyde (MDA) cause lipid peroxidation. (9) It is among the information in the literature that MDA levels increase in the case of periodontal inflammation and that MDA can be considered as an oxidative stress marker for periodontitis. (10-12)
glutathione | 1 year
  Glutathione (GSH) acts as a coenzyme in the oxidation-reduction process. (15) GSH is a critical redox regulator and important for the health of peridontium

CONTACTS AND LOCATIONS:
Overall Officials: hacer sahin aydınyurtt, assoc. prof, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van yuzuncu yil university, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided